CLINICAL TRIAL: NCT03052348
Title: A Multicentre Study Evaluating the Efficacy of Combining Topical Antibiotic/Steroid/Moisturizer Therapy Compared to Standard of Care in the Treatment of Severe Atopic Dermatitis, a Phase II Randomized, Clinical Trial
Brief Title: Efficacy of Combining Topical Antibiotic/Steroid/Moisturizer Therapy Compared to Active Comparator in Atopic Dermatitis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Red Cross War Memorial Childrens Hospital (Other)
Responsible Party: Principal Investigator, Dr Carol Hlela, Dr, Red Cross War Memorial Childrens Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RedCrossWMCH
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Severe Atopic Dermatitis
Keywords: Topical Antibiotics; Fusidic Acid; Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Cetomacrogol; Fusidic Acid

STUDY DESIGN:
Intervention Model Description: Fusidic acid, polyethylene glycol hexadecyl ether & Betamethasone valerate cream 0.1%
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be given creams (containing either the intervention or control regimens - both white in color) in unlabelled opaque containers. Participants, investigators and the outcomes assessor evaluating the outcome of interest (SCORAD) will be blinded to the treatment allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group R (Active Comparator): Polyethylene glycol hexadecyl ether & betamethasone valerate cream 0.1% . ( 4 applications per day for 14 days treatment to taper fortnightly)
  Interventions: Other: Polyethylene glycol hexadecyl ether & Betamethasone valerate cream 0.1%
- Group A (Experimental): Fusidic acid & Polyethylene glycol hexadecyl ether,& betamethasone valerate cream 0.1%). ( 4 applications per day for 14 days treatment to taper fortnightly)
  Interventions: Other: Fusidic acid, polyethylene glycol hexadecyl ether & Betamethasone valerate cream 0.1%

INTERVENTIONS:
Other: Polyethylene glycol hexadecyl ether & Betamethasone valerate cream 0.1% — Polyethylene glycol hexadecyl ether -Moisturizer. Betamethasone valerate cream 0.1% -Topical steroid
  Other Names: Cetomacrogol 400g, Reg No PL 00240/0014.; Lenovate cream, 15g, Reg No. 27/13.4.1/0493
  Arms: Group R
Other: Fusidic acid, polyethylene glycol hexadecyl ether & Betamethasone valerate cream 0.1% — Polyethylene glycol hexadecyl ether -Moisturizer. Betamethasone valerate cream 0.1% -Topical steroid Fusidic Acid - Topical Antibiotic
  Other Names: Cetomacrogol 400g, Reg No PL 00240/0014.; Lenovate cream, 15g, Reg No. 27/13.4.1/0493; Fusidic Acid (Fucidin cream), 15 g, Reg No. Q/20.1.6/128
  Arms: Group A

SUMMARY:
Atopic dermatitis (AD) is a chronic, relapsing inflammatory skin disease that occurs most commonly during early infancy and childhood. It is frequently associated with abnormalities in skin barrier function, allergen sensitization and recurrent skin infections. AD is a major public health problem worldwide, with prevalence in children of 10-20% and 2-5% of the general population. The skin of AD patients is susceptible to colonization and infection with Staphylococcus aureus (SA )which contribute significantly to the severity of the clinical manifestations of eczema, triggering a vicious cycle.

Fusidic Acid (FA) cream is a topical antibiotic widely used in the treatment of skin and soft tissue infections and infected atopic dermatitis. However in recent years, the emergence of drug-resistant organisms, e.g. Methicillin- resistant Staphylococcus aureus (MRSA) has led to scrutiny of antibiotic use. Prolonged use of topical FA has been linked with emergence of FA-resistant Staphylococcus aureus (FRSA) . Fusidic acid is a natural antibiotic, extracted from cultures of Fusidium coccineum, which has a powerful antibacterial action. Topical use of Fusidic acid is fully in line with therapeutic strategies that recommend the use of an antibiotic with the narrowest activity spectrum to minimize the risk of resistance. In AD with infected lesions, combined treatment with antibiotic and steroid demonstrates greater efficacy over the use of steroid.

Trial Design: A three-center, double blind, randomized ,phase II , parallel group, efficacy trial.

Type of Intervention: A triple compounded cream containing a topical antibiotic , topical steroid and moisturizer.

Type of control: Active control containing a double compounded cream comprising a topical steroid and moisturizer .

Study population and Setting: A sample of 78 subjects will be recruited from Red Cross Children's Hospital , Nelson Mandela Academic Hospital and King Edward Hospital Estimated duration of trial: 12 months. Duration of participation: Each subject will participate in the trial for a maximum of 140 days.

Primary endpoint: reduction in SCORAD scores; frequency of clinical flares for AD and improvement in the quality of life at 140 days.

The benefit of this trial is that it provides a simple and effective approach to the management of atopic eczema.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a parent/legally authorized representative, who is able to give informed consent and willing and able to comply with all the required study procedures. Assent is required from children who in the investigator's judgement, are capable of understanding the nature of the study.
* Participants must have have AD as defined by the UK Working Party Criteria
* Participants can be female or male, older than 2 years but younger than 10 years (up to their 10th birthday)
* Participants must not be on systemic antibiotics treatment at recruitment
* Participants must have a baseline SCORAD score of 50 or above (severe AD)
* Participants must be eligible for second line treatment agents for AD (systemic or photo therapy)

Exclusion Criteria:

* Participants must not be systemic agents (e.g. immunosuppressive) for AD
* Participants must not be younger than 2 years or over 10 years in age.
* Participants must not be using g bleach baths as a staphylococcus eradication measure at the time of enrollment,
* Participants must not have mild-moderate AD (SCORAD< 50)
* Participants must not be immune-compromised with AD
* Participants must not be on photo therapy for AD
* Participants must not be using wet wrap therapy for AD

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-08-30 (Estimated)

PRIMARY OUTCOMES:
SCORAD scores | 20 weeks
  Reduction of SCORAD scores in the treatment group (A) of patients comparing with scores in the control group (R), at the end of the study with reference to baseline

SECONDARY OUTCOMES:
Infants Dermatitis' Quality of Life (IDQOL) index | 20 weeks
  Improvement in the Infants Dermatitis' Quality of Life (IDQOL) index in group (A) patients compared to that of the control group (R) at the end of the study compared to baseline
Frequency of AD relapse episodes | 20 Weeks
  Comparison of the frequency of AD relapse episodes in group (A) patients compared to the frequency of relapse episodes in control group (R) patients.
Time to AD Relapse | 20 weeks
  Comparison of the time to AD relapse episodes in group (A) patients compared to the time to relapse episodes in control group (R) patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Carol Hlela, MBCHB, Principal Investigator — Red Cross Children's War Memorial Hospital
Locations (3):
- South Africa (3):
  - Nelson Mandela Academic Hospital, Mthatha, Eastern Cape
  - King Edward Hospital, Durban, KwaZulu-Natal
  - Red Cross War Memorial Children's Hospital, Cape Town, Western Cape

REFERENCES:
- [Background] Sidbury R, Tom WL, Bergman JN, Cooper KD, Silverman RA, Berger TG, Chamlin SL, Cohen DE, Cordoro KM, Davis DM, Feldman SR, Hanifin JM, Krol A, Margolis DJ, Paller AS, Schwarzenberger K, Simpson EL, Williams HC, Elmets CA, Block J, Harrod CG, Smith Begolka W, Eichenfield LF. Guidelines of care for the management of atopic dermatitis: Section 4. Prevention of disease flares and use of adjunctive therapies and approaches. J Am Acad Dermatol. 2014 Dec;71(6):1218-33. doi: 10.1016/j.jaad.2014.08.038. Epub 2014 Sep 26. PMID 25264237
- [Background] Cardona ID, Cho SH, Leung DY. Role of bacterial superantigens in atopic dermatitis : implications for future therapeutic strategies. Am J Clin Dermatol. 2006;7(5):273-9. doi: 10.2165/00128071-200607050-00001. PMID 17007538
- [Background] Huang JT, Abrams M, Tlougan B, Rademaker A, Paller AS. Treatment of Staphylococcus aureus colonization in atopic dermatitis decreases disease severity. Pediatrics. 2009 May;123(5):e808-14. doi: 10.1542/peds.2008-2217. PMID 19403473
- [Background] Langan SM, Thomas KS, Williams HC. What is meant by a "flare" in atopic dermatitis? A systematic review and proposal. Arch Dermatol. 2006 Sep;142(9):1190-6. doi: 10.1001/archderm.142.9.1190. PMID 16983006
- [Background] Totte JE, van der Feltz WT, Hennekam M, van Belkum A, van Zuuren EJ, Pasmans SG. Prevalence and odds of Staphylococcus aureus carriage in atopic dermatitis: a systematic review and meta-analysis. Br J Dermatol. 2016 Oct;175(4):687-95. doi: 10.1111/bjd.14566. Epub 2016 Jul 5. PMID 26994362
- [Background] Nakamura Y, Oscherwitz J, Cease KB, Chan SM, Munoz-Planillo R, Hasegawa M, Villaruz AE, Cheung GY, McGavin MJ, Travers JB, Otto M, Inohara N, Nunez G. Staphylococcus delta-toxin induces allergic skin disease by activating mast cells. Nature. 2013 Nov 21;503(7476):397-401. doi: 10.1038/nature12655. Epub 2013 Oct 30. PMID 24172897